CLINICAL TRIAL: NCT04097080
Title: Comparative Controlled Study of Analgesic, Antiasthenic and Anti-Anxiety Effects of Xenon in Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nobilis Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBTX-009
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBTX-001 (Experimental): 30% medical grade xenon/70% Oxygen
  Interventions: Drug: NBTX-001
- Standard of Care (Placebo Comparator): Reconstituted air
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: NBTX-001 — Active drug group will receive 6 doses of NBTX-001 given three times a week.
  Arms: NBTX-001
Drug: Standard of Care — Placebo group will receive reconstituted air given three times a week.
  Arms: Standard of Care

SUMMARY:
This study evaluates the hypothesis that the gas mixture with xenon will have a positive effect on the symptoms in patients with Parkinson's Disease. The study will test the hypothesis that the gas mixture with xenon has a symptomatic treatment potential for patients with Parkinson's Disease, as measured by change from baseline in the Unified Parkinson Disease Rating Scale (UPDRS).

ELIGIBILITY:
Inclusion Criteria:

* The patient must be male or female over the age of 18.
* The subject must have idiopathic Parkinson's disease.
* The subject has Stage III by Hoehn and Yahr in the "on" state on a screening visit
* Subjects suffering from anxiety, depression, cognitive dysfunction
* Dopaminergic drugs should be taken in a stable dosage for 28 days prior to registration, and throughout the study
* Patients who have signed an approved consent form and are consistent with both the clinical trial plan and follow-up.

Exclusion Criteria:

* Patients have atypical parkinsonism (eg, neuroleptics, metoclopramide, flunarizin), metabolic neurodegenerative disorders (eg, Wilson's disease), encephalitis, cerebrovascular disease or degenerative disease (e.g. progressive supranuclear palsy)
* Patients who received deep brain stimulation
* Patients with cancer, HIV, kidney or liver disease.
* Patients taking new antipsychotic, antidepressant, anxiolytic or narcotic drugs for less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson Disease Rating Scale (UPDRS) | Baseline to Week 24
  Analysis of Unified Parkinson Disease Rating Scale (UPDRS) from baseline.The UPDRS scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients. The UPDRS scale includes series of ratings for typical Parkinson's symptoms that cover all of the movement hindrances of Parkinson's disease. The UPDRS scale consists of the following five segments: 1) Mentation, Behavior, and Mood, 2) ADL, 3) Motor sections, 4) Modified Hoehn and Yahr Scale, and 5) Schwab and England ADL scale. Each answer to the scale is evaluated by a medical professional that specializes in Parkinson's disease during patient interviews. Some sections of the UPDRS scale require multiple grades assigned to each extremity with a possible maximum of 199 points. A score of 199 on the UPDRS scale represents the worst (total disability) with a score of zero representing (no disability).

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Institute of Addictology, Moscow
  - MONIKI, Moscow